CLINICAL TRIAL: NCT02053818
Title: Fast-track in Cardiac Surgery. Remifentanyl & Sufentanil Anaesthesia for CABG+/-AVR Evaluated by Recovery, Cognitive Dysfunction, Haemodynamics (PAC/TTE) and Cardiac Biochemical Markers (CKMB, TNT, Pro-BNP)
Brief Title: Remifentanil/Sufentanil for CABG+/-AVR Evaluated by Recovery, Cognitive Function, Haemodynamics and Biochemical Markers.
Acronym: PRECON2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Carl-Johan Jakobsen, Research Consultant, Ass professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-022428-58
Record Dates: First submitted 2014-01-06; First posted 2014-02-04 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Ischaemic Heart Disease; Aortic Stenosis
Keywords: Cognitive dysfunction; Cardioprotection; Recovery; Renal function; ICU discharge
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis; Cognitive Dysfunction | interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Active Comparator): Remifentanil the basic opioid drug in anesthesia
  Interventions: Drug: Remifentanil
- Sufentanil (Active Comparator): Sufentanil the basic opioid drug in anesthesia
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Remifentanil — Randomization to receive Remifentanil (ultrashort acting opioid) as basic opioid in anaesthesia
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Sufentanil — Randomization to receive Sufentanil (medium/long acting opioid) as basic opioid in anaesthesia
  Other Names: Sufenta
  Arms: Sufentanil

SUMMARY:
To evaluate the effect on cognitive function, recovery, cardioprotection and haemodynamics of standard Remifentanil anaesthesia to standard Sufentanil anaesthesia in patients undergoing coronary artery bypass with or without aortic valve replacement.

DETAILED DESCRIPTION:
1. Haemodynamic effects, evaluated by invasive haemodynamic data (arterial line and PAC) of opioid given as single drug and in combination with Propofol (first 30 patients only).
2. Cognitive dysfunction evaluated by standard test preoperative and postoperative day 1, 4 and 30
3. Recovery quality and time parameters using objective ICU score criteria
4. Cardioprotection effect evaluated by myocardial biochemical markers obtained preoperative and postoperative 4, 9 and 18 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for coronary artery bypass grafting (CABG) +/- aortic valve replacement (AVR)

Exclusion Criteria:

* Ejection Fraction < 30%
* Previous Myocardial Infarction within 4 weeks
* Severe pulmonary hypertension (mean pulmonary artery pressure (mPAP) > 33% of mean arterial pressure (MAP)
* Arterial hypertension (Sap > 180, Dap > 110)
* Diabetes, Non- and Insulin dependent
* Non usable echocardiography windows

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Cognitive function score | Postoperative day 4
  Cognitive function evaluated by Palo Alto Veterans Hospital Test on all patients
Fast-track potential | Time ((mean hours) to eligible discharge from ICU (up to 48 hours)
  Ventilation time and eligible time to discharge based on ICU score

SECONDARY OUTCOMES:
Eligible time to discharge from ICU | Time (hours) to ICD4
  Estimation on hours in ICU before the patients were eligible for discharge from ICU = ICD4 (Total score < 5, and no single score > 2) using an objective ICU score. The ICU score is done each hour after extubation
Postoperative cognitive dysfunction | Postoperative day 1 and 30
  Changes from pre-operative cognitive function to postoperative cognitive function on day 1, 4 and 30 using cognitive function test from Palo Alto Veterans Hospital Test on all patients

OTHER OUTCOMES:
Haemodynamic effects of opioids | From induction anaesthesia until cardiopulmonary bypass
  Evaluation of haemodynamic indexes (cardiac index, stroke volume index, central venous oxygenation, blood pressure, Heart rate) together with echocardiographic evaluation of systolic and diastolic function.
  Evaluation both by single opioid and combination with propofol
Cardioprotection | 0,4,9,15 and 40 hours after surgery
  Evaluation based on myocardial biochemical markers CK-MB, Troponin-T and Nt-Pro-BNP preoperative and 4, 9 and 15 and 40 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Johan Jakobsen, MD, Study Director — Department of Anaesthesiology and Intensive Care, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark